CLINICAL TRIAL: NCT03712527
Title: A Randomized, Double-blind Controlled Trial of the Efficacy of an Intra-discal Injection of Autologous Platelet-rich Plasma (PRP) Versus Placebo in Chronic Low Back Pain With Active Discopathy (AD)
Brief Title: Intra-discal Injection of PRP for Low Back Pain
Acronym: MODI-PRP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL18_0036; 2018-000872-14 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-07-23; First posted 2018-10-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain
Keywords: Active discopathy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet-Rich Plasma (Experimental)
  Interventions: Other: Injection of Platelet rich plasma
- Placebo (Placebo Comparator)
  Interventions: Other: Injection of NaCl

INTERVENTIONS:
Other: Injection of Platelet rich plasma — The blood of the PRP patients group will be centrifuged by the nurse using the dedicated device. A single centrifugation is required to separate the red and white blood platelets and plasma. This method of centrifugation is carried out using specific kits (Mini-GPS System III, Zimmer Biomet Company). The PRP is then collected by the nurse into a syringe that will be provided to the injector physician. Duration of preparation: 20 to 25 minutes. After a standardized sterile preparation, a local anaesthesia will be performed. Then, the injector will inject a volume of 2 mL of PRP into the median portion of the suspected disc under radiographic guidance.
  Arms: Platelet-Rich Plasma
Other: Injection of NaCl — The placebo will be a single-dose of saline solution which corresponds to NaCl 0,9% ProAmp 10 ml (Laboratoire Aguettant). The vials will be kept at room temperature (≤ 25°C) within the local pharmacy of each centre. 2 mL of this solution will be intra-discal injected.
  Arms: Placebo

SUMMARY:
Low back pain (LBP) is the second cause of medical visits in France. Indeed, its incidence can vary between 60 and 90%. LBP is also the leading cause of disability in the adult population in France and in the rest of the world. Its evolution towards chronicity is observed in less than 8% of cases, but it is responsible for 85% of the medical costs. Degenerative disk disease (DDD) is a major cause of chronic LBP (> 40%). DDD can be characterized by peculiar Magnetic Resonance Imaging (MRI) features with a strong correlation between pain and inflammatory aspect of the disk, which result in the so-called active discopathy (AD) (Brinjikji et al. 2015). Modic classification based on MRI of the lumbar spine is considered as a reference. Type 1 Modic signal changes are characterised by a low-intensity signal on T1-weighted sequences and hyperintense signal on T2-weighted sequences, with gadolinium injection enhancement, corresponding to bone marrow oedema. Type 1 Modic is very rare in an asymptomatic population but may be found in 5% to 40% of chronic LBP patients underscoring its symptomatic involvement. No currently reference treatment is available for AD.

PRP technology has recently been widely developed in osteoarthritis and tendon injuries. Therapeutic benefit of PRP has being evaluated. For instance, no randomized controlled trials (RCTs) have specifically evaluated the effect of PRP in AD (Modic 1 signal). The availability of PRP for intra- discal injection could become an innovative therapeutic option in humans, especially for AD forms where inflammatory process is clearly predominant.

The objective of the study is to evaluate the 3-month efficacy on pain and function (by achieving 30% improvement in Oswestry Disability Index) of one intra-discal PRP injection versus placebo (saline solution) in subjects with LBP associated with AD lasting more than 3 months.

ELIGIBILITY:
Inclusion Criteria:

* - Age between 18 to 60 years
* Patient with AD characterized by a common lumbar spine for more than 3 months associated with Modic I discopathy on MRI on a single level
* Annulus fibrosus capable of holding the cell implantation, demonstrated by MRI (stages < 5 of Pfirrmann's score). The Pfirrmann's score is fully described in annex (Pfirrmann et al. 2001).
* Daily LBP for at least 3 month with baseline mean intensity ≥ 40 mm on VAS (0-100) in the previous 48 hours
* Written and signed informed consent form
* Subjects must be covered by public health insurance
* Subjects must be able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* - Patient with Modic 1 discopathy in different vertebral levels
* Patient with a Modic I signal abnormality related to a static spinal disorder (such as previous vertebral fractures, or isthmic lysis, or spondyloarthritis)
* Patient with a history of lumbar spine surgery
* Patient with suspected spondylodiscitis or other infection
* Patient under anticoagulant or antiaggregant therapy, or with a coagulation disorder
* Patient with allergy to iodine or to any of the components of Xylocaine
* Contraindication to MRI: Pacemaker or neurosensorial stimulator or implantable defibrillator, cochlear implant, ferromagnetic foreign body similar to the nervous structure.
* Patient with anatomical difficulty of access to the injection area (judged by the investigator)
* Patient with an uncontrolled severe disease (i.e. heart, pulmonary, gastro-intestinal, neurologic, endocrine, auto-immune affections) limiting the patient's safety (judged by the investigator)
* Patient with previous malignancy less than 5 years (except for non-melanoma skin cancer)
* Prior to the screening visit:
* a current and recent use of morphine (< 1 month)
* a systemic or local corticosteroid therapy (< 1 month)
* Porphyria
* Patient with sphincter disorders indicating a cauda equina syndrome
* Psychotic state not controlled by a treatment
* Pregnancy (βHCG positive), breast-feeding or the absence of effective contraception for women of child-bearing age
* Vulnerable persons protected by law
* Persons under guardianship
* Subject who are in a dependency or employment with the sponsor or the investigator
* Participation in another clinical trial
* Subject unable to read or/and write

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the functional disability | Baseline, 3 months
  The Oswestry Disability Index is a questionnary used to evaluate functional disability. A patient is considered as responder if he/she manages to achieve at least 30% improvement in this score between baseline and 3 months. This self-completed questionnaire contains ten topics concerning intensity of pain, and activities of daily life. Each topic category contains 6 statements describing a growing degree of relative severity to a particular activity. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 where zero indicates the least amount of disability and 5 indicating most severe disability. The ODI scale range from 0 to 100 where zero corresponds to no disability and 100 is the maximum disability possible. The ODI minimum detectable change is 10% points. That means at least a 10% change is required to be clinically meaningful.

SECONDARY OUTCOMES:
Disability evaluation (RMQ questionnaire) | Baseline, 1, 3, 6 and 12 months
  Functionnal disability will be assessed by the Roland Morris Questionnaire (RMQ). RMQ is a 24-item self-report questionnaire designed to assess physical disability and functional limitations caused by LBP. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability). For the RMQ, a between-groups difference of 2 points is considered clinically important, whereas a within-patient change of 4 or 5 points is recognized as the threshold for a clinically important improvement.
Disability evaluation (MCID) | Baseline,1,3 and 6 months
  The minimal clinically important difference (MCID). MCID reflects the concept of improvement ("feeling better"). The patient acceptable symptom state (PASS) has been proposed to address the concept of partial symptomatic remission ("feeling good"). The concept of the MCID defines the smallest meaningful change score for outcome measures.Published MCID values for the included instruments range from 15 of 100 for absolute improvement (MCID).
Disability evaluation (PASS) | Baseline,1,3 and 6 months
  The Patient acceptable symptomatic state (PASS) has been proposed to address the concept of partial symptomatic remission ("feeling good"). The PASS value is a clinically relevant cutoff from the patient's perspective, which allows for classifying patients at the end of the trial as being in "an acceptable state" (with the outcome score ≤ the PASS) or not (with the outcome score > the PASS). Published MCID and PASS values for the included instruments range from 40 of 100 (PASS).
Assessment of pain and conséquences (Efficacy) | Baseline, 1, 3, 6 and 12 months
  Visual analogue scale (VAS), use of analgesics and Non steroidal anti inflammatory drugs (NSAIDs). Scale used to assess pain. Measurement of pain killer drugs
Assessment of pain and conséquences (Employement and work status) | Baseline, 1, 3, 6 and 12 months
  Employment and work status will be assessed. For this we will assign each of the patients to one of 4 categories designated as "employable" which included those who were unemployed due to pain, employed but on sick leave, laid off, or working. The other categories include retired, disabled, and elderly at least 60 years of age, eligible for social security. The number of days of work absence will be recorded during each follow-up visit. The resumption of professional activity will be requested to the patient at each visit. The type of resumption will be notified. A return to the patient's employment or a prolonged work stoppage are expected as a result.
The number of consumption of analgesics | Baseline, 1, 3, 6 and 12 months
  The analgesic consumption will be analysed in order to show a change of the analgesic consumption.The use of analgesics will be registered on a patient booklet with weekly collection.
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | Baseline, 1, 3, 6 and 12 months
  measurement of safety along the study Adverse events, incidence, relatedness, severity of treatement-emergent SUSARs, SAEs, Ars and AEs
Changes in quality of life, EQ5D questionnaire (Efficacy) | Baseline, 1, 3, 6 and 12 months
  EQ-5D is a standardized instrument developed as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments.This score varies between 0 and 1: 0 represents death, and 1 the best quality of life possible. So, this score indicates the decrease in quality of life compared to an optimal state of health. The more desirable a health state, the higher the score associated with it. Negative scores are possible if the subject perceives a state of health worse than death. The EQ-5D includes the following five dimensions: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression.
Changes in quality of life, SF36 questionnaire (Efficacy) | Baseline, 1, 3, 6 and 12 months
  The SF-36 includes 36 items divided into 8 dimensions (physical functioning, limitations of functions related to physical health, physical pain, general health, vitality [energy / fatigue], functioning or social well-being, limitations of functions related to mental health, physical health) to which were added 4 items examining the cognitive functioning, from the "Medical Outcomes Study". This questionnaire was supplemented by questions aimed at clarifying the socio-demographic profile of the participants as well as the use of care services.

CONTACTS AND LOCATIONS:
Overall Officials: Yves-Marie PERS, Principal Investigator — University Hospital, Montpellier
Locations (6):
- France (6):
  - CHU Bordeaux, Bordeaux
  - Univesity Hospital od Montpellier, Montpellier
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - APHP Cochin, Paris
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided